CLINICAL TRIAL: NCT07051798
Title: Phlebitis Experiences of Intensive Care Nurses: A Qualitative Study
Brief Title: Phlebitis Experiences of Intensive Care Nurses
Status: Recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Sponsor
Other Study IDs: KHSU20250607
Record Dates: First submitted 2025-06-12; First posted 2025-07-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Phlebitis; NursİNG CARE
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: It is a qualitative type of study that will be conducted through face-to-face interviews. — It is a qualitative type of study that will be conducted through face-to-face interviews.

SUMMARY:
It is important to reveal the phlebitis experiences of nurses. The data obtained from the phlebitis experiences of nurses are important in terms of preventing phlebitis and supporting patient safety practices. In the studies conducted to date, no study has been found in the literature that qualitatively examines the phlebitis experiences of intensive care nurses. This study is the first to be conducted in this respect, which constitutes the originality of the research. It is expected to guide clinician and academic nurses in phlebitis assessment and phlebitis care planning and to contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily accepting to participate in the study
* Being the primary nurse of a patient who developed phlebitis,
* Having at least 1 year of work experience.

Exclusion Criteria:

* Being assigned to the unit for a short period of time
* Being on leave or sick leave,
* Not accepting to participate in the study,
* Leaving the study during the data collection process.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Intensive Care nurses
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Themes Identified in ICU Nurses' Experiences with Phlebitis Management | Within the first 2 months following the initiation of the study
  Identification of distinct thematic categories from ICU nurses' experiences concerning the recognition, prevention, care practices, and clinical challenges related to phlebitis. Each theme will be extracted through thematic analysis of qualitative data obtained from semi-structured interviews. Method of Analysis: Braun & Clarke's Thematic Analysis Method Unit of Measure: Number of distinct themes identified
Perceived Barriers and Facilitators in Phlebitis Management | Within 2 month after the completion of data collection
  Evaluation and classification of ICU nurses' perceptions regarding institutional, educational, and individual-level factors affecting phlebitis assessment and management. Each perceived barrier or facilitator will be categorized based on content analysis of semi-structured interview transcripts. Method of Analysis: Content Analysis Methodology Unit of Measure: Number of identified barriers and facilitators.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No